CLINICAL TRIAL: NCT01652027
Title: Study of Immunologic Determinants of Inhibitor Development in Previously Untreated Patients With Hemophilia
Brief Title: Hemophilia Inhibitor Previously Untreated Patient Study
Acronym: HIPS
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Rho, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Deborah Brown, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-11-0202; HSC-MS-11-0202 (Other: University of Texas HSC-Houston Committee for the Protection of Human Subjects)
Record Dates: First submitted 2011-06-03; First posted 2012-07-27 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Hemophilia A
Keywords: FVIII inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples, lymphocyte cell lines, Genomic DNA, RNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Previously Untreated Patients with Hemophilia A
  Interventions: Drug: FVIII concentrate

INTERVENTIONS:
Drug: FVIII concentrate — usual treatment as directed by treating physician

SUMMARY:
Hemophilia A is a congenital bleeding disorder caused by deficiency of factor VIII (FVIII) and is treated by replacement therapy with FVIII concentrate. Approximately 30% of people with severe hemophilia A develop neutralizing antibodies, called FVIII inhibitors, which interfere with the function of FVIII concentrates. The reason that some, but not all, people with severe hemophilia A develop inhibitors is incompletely understood. Understanding individual and environmental risk factors is important to be able to prevent and possibly treat inhibitors. This study will look at individual and treatment characteristics in babies with severe hemophilia A who have not yet received treatment with FVIII (called Previously Untreated Patients, or PUPS). Subjects in the study will be asked to provide diaries of treatments, medications, and illnesses. Treatment will be directed by the subjects' physician, but all subjects will receive Advate, a third-generation recombinant FVIII product. Subjects will have blood drawn for laboratory tests, which include studies of the immune system and genetic studies of the FVIII mutation, before and 7-9 days after the first treatment with FVIII, and 5 days (+/-2 days) after the 5th, 10th, 20th, 30th, 40th, and 50th days of treatment with FVIII (exposure days). The duration of the study will be first 50 treatments or 3 years, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A with FVIII activity < 1% normal
* Weight > 3.5 kg at the time of baseline study evaluation
* Informed consent, approved by appropriate Institutional Review Board/Independent Ethics Committee, has been administered, signed, and dated

Exclusion Criteria:

* Prior exposure to clotting factor concentrates or blood products
* Other chronic disease
* Currently participating in another investigational drug study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe hemophilia A who have not previously been treated with Factor VIII concentrates.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Total number of FOXP3-positive T regulatory cells in the circulation | 50 exposure days to FVIII or 3 years, whichever comes first
  FoxP3(a protein involved in immune system responses)-positive T regulatory cells in the circulation will be compared before and after exposure to FVIII.

SECONDARY OUTCOMES:
FVIII-specific T-cells | 50 exposure days to FVIII or 3 years, whichever comes first
  FVIII-specific T-cells will be compared before and after exposure to FVIII

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, M.D., Principal Investigator — Maggiore Hospital and University of Milan
Locations (17):
- United States (13):
  - Emory University, Atlanta, Georgia
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Cornell University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Oregon, Portland, Oregon
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - North Texas Comprehensive Hemophilia Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center-Houston, Houston, Texas
  - Intermountain Hemophilia and Thrombosis Center, Salt Lake City, Utah
- Medical University of Vienna, Vienna, Austria
- Angelo Bianchi Bonomi Hemophilia & Thrombosis Center, Milan, Italy
- Emma Children's Hospital AMC, Amsterdam, Netherlands
- Malmo Centre for Thrombosis and Haemostasis, Malmo, Sweden

REFERENCES:
- [Derived] Paul H, Berg V, Gangadharan B, Bowen J, LeBeau P, Blatny J, Male C, Radulescu VC, Diaz R, Mancuso ME, Brown DL, Reipert BM. Prospective Hemophilia Inhibitor PUP Study reveals distinct antibody signatures during FVIII inhibitor eradication. Blood Adv. 2023 May 9;7(9):1831-1848. doi: 10.1182/bloodadvances.2022007267. PMID 36074992
- [Derived] Reipert BM, Gangadharan B, Hofbauer CJ, Berg V, Schweiger H, Bowen J, Blatny J, Fijnvandraat K, Mullins ES, Klintman J, Male C, McGuinn C, Meeks SL, Radulescu VC, Ragni MV, Recht M, Shapiro AD, Staber JM, Yaish HM, Santagostino E, Brown DL. The prospective Hemophilia Inhibitor PUP Study reveals distinct antibody signatures prior to FVIII inhibitor development. Blood Adv. 2020 Nov 24;4(22):5785-5796. doi: 10.1182/bloodadvances.2020002731. PMID 33232473